CLINICAL TRIAL: NCT06047509
Title: Focal Laser Ablation of Prostate Cancer: A Feasibility Study Using MRI/US Image Fusion for Guidance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-001942
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: the investigators intend to use Focal Laser Ablation guided by the UnfoldAI software to identify cancer margins and create ablation treatment plans and use the FocalPoint System to deploy and monitor thermal energy in cancerous regions of the prostate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm I Treatment (Experimental): After inserting the laser, a thermal-optical probe will be inserted via a multichannel needle guide or tranperineal grid in the prostate using transrectal ultrasound guidance. The sensor probe will be placed at a pre-determined depth and location based on the treatment zone. Targets will be identified prior to laser treatment using multi-parametric MRI and delineated by the radiologist for visualization by the treatment operator. The lesion will be visible both on a 3D reconstruction and during real-time ultrasound imaging. Applications of laser energy up to 15 watts of power will be used to treat the target region. Confirmation of appropriate laser position will be made with real-time ultrasound prior to application of laser energy and repeatedly during activation of the laser. Energy delivery will be planned specific to each patient's tumor geometry, with the assistance of the Avenda Health Unfold-AI Software.
  Interventions: Procedure: Focal Laser Ablation

INTERVENTIONS:
Procedure: Focal Laser Ablation — Removal of cancerous tissue through the direct application of laser energy
  Other Names: FLA

SUMMARY:
This is an open-label feasibility/pilot study to evaluate the safety and feasibility of the FocalPoint System with UnfoldAI. In this study, the investigators intend to use the UnfoldAI software to identify cancer margins and create ablation treatment plans and use the FocalPoint System to deploy and monitor thermal energy in cancerous regions of the prostate. Subjects will be assessed at 1 week, 1 month, and every 3 months until one-year post-FLA treatment(s) to be monitored for adverse events and complete quality-of-life questionnaires.

DETAILED DESCRIPTION:
The Avenda Health FocalPoint System (K201687) is a laser-based interstitial irradiation/thermal soft-tissue ablation system that is FDA 510(k) cleared for surgical applications requiring the vaporization, incision, excision, ablation, cutting and hemostasis, or coagulation of soft tissue in conjunction with endoscopic equipment for various medical specialties. The Avenda Health Unfold-AI Software (K221624) is an Artificial Intelligence (AI)-based decision support software, indicated as an adjunct to the review of magnetic resonance (MR) prostate images and biopsy findings in the prostate oncological workflow that is also FDA 510(k) cleared. The Unfold-AI Software will be utilized along with the FocalPoint System and is designed to support the prostate oncological workflow by helping the user with the segmentation of MR image features, including the prostate; in the evaluation, quantification, and documentation of lesions; and in pre-planning for diagnostic and interventional procedures such as biopsy and/or soft tissue ablation. This feasibility investigation will determine whether the FocalPoint System used with Unfold-AI can be used to ablate prostate tissue in men with prostate cancer while leaving critical structures (urethra, rectal wall) undamaged.

This is an open-label feasibility/pilot study to evaluate the safety and feasibility of the FocalPoint System with Unfold-AI. In this study, the investigators intend to use the Unfold-AI software to identify cancer margins and create ablation treatment plans and use the FocalPoint System to deploy and monitor thermal energy in cancerous regions of the prostate. MRI guidance will be achieved by MRI/ultrasound fusion, overlaying stored MRI images upon real-time ultrasound images. Interstitial laser treatments would be achieved by inserting the fiber into the cancerous regions guided by the Artemis image-fusion device. Applications of laser energy up to 15 watts of power will be used to treat the target region. Subjects will be assessed at 1 week, 1 month, and every 3 months until one-year post-FLA treatment(s) to be monitored for adverse events and complete HRQOL questionnaires. Post-treatment MRI findings, fusion biopsy results and biomarker (PSA) kinetics will also be monitored. Subjects eligible for repeat FLA (re-ablation) are those who still continue to meet Inclusion and Exclusion Criteria at Months 6 or 12 post-FLA treatment (See Sections 3.0 Inclusion Criteria, 4.0 Exclusion Criteria, and 6.4.7 Repeat FLA (re-ablation)). Subjects may undergo only one re-ablation on the study.

This study will cover pre-treatment through 12 months following FLA treatment or repeat FLA (re-ablation) treatment. The study also has a long-term follow-up data collection period of up to 10 years following a subject's last study visit.

The primary endpoint will be safety. Safety will be determined by the number, type, and severity of adverse events incurred by subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with organ-confined prostate cancer (clinical stage ≤ T2b, Gleason =7)
* Age 40 to 85 years of age
* Multi-parametric MRI read at study site within 9 months of study treatment, demonstrating a Region of interest (ROI) of MRI (PIRADSv2 > Grade 3)1
* Prostate volume 20cc to 80cc
* MRI/ultrasound fusion biopsy with ≥ 10 systematic biopsy cores and ≥ 2 targeted biopsy cores from above MRI-derived ROI within 6 months of study treatment*
* Histologically confirmed adenocarcinoma from targeted biopsy cores
* Overall Gleason = 3+4 or 4+3
* Subjects desire focal therapy and decline conventional treatment (active surveillance, radical prostatectomy, radiation therapy, cryosurgery, and hormone therapy)
* Treatment plan that allows for treatment of lesion while still maintaining a 4mm safety margin from the rectal wall and urethra
* Signed informed consent for the FLA treatment through follow-up per study protocol

  * For subjects under consideration for repeat FLA, the post-treatment MRI and biopsies done at Months 6 and 12 study visits may be used for these criteria.

Exclusion Criteria:

* Any significant cancer outside of the intended treatment zone, defined as Gleason score ≥ 7
* < 10 years life expectancy
* Any medical condition that would compromise the subject's ability to safely participate in the study
* Active bleeding disorder
* Use of coumadin or any other anticoagulant, unless anticoagulation can be temporarily reversed or stopped for a window of at least 7 days peri-procedure
* Use of aspirin, unless it can be temporarily stopped for a window of at least 14 days prior to FLA procedure
* Use of NSAIDS (except aspirin), Vitamin E, multivitamins, and herbal products, unless they can be temporarily stopped for at least 7 days prior to FLA procedure
* Active urinary tract infection
* Active prostate abscess, prostatitis, or neurogenic bladder
* Any prior treatment for prostate cancer, including:

  * Radical prostatectomy
  * Radiation therapy (external beam or brachytherapy)
  * Cryotherapy
  * High intensity focused ultrasound (HIFU) treatment
  * Photodynamic therapy
  * Androgen deprivation therapy
  * Focal Laser Ablation (acceptable for enrolled subjects under consideration for repeat FLA)
* Prior prostate, bladder neck, or urethral stricture surgery
* Any prostate debulking procedure, including transurethral resection of prostate, photovaporization, or electrovaporization
* Transurethral incision of bladder neck
* Urethral stricture dilation or reconstruction
* Use of 5-alpha reductase inhibitors within 6 months of treatment
* Prior significant rectal surgery (hemorrhoidectomy is acceptable)
* Active rectal fissure, fibrosis, stenosis, or other anatomic abnormality precluding insertion of transrectal device
* Active inflammatory bowel disease
* Urinary tract or rectal fistula
* Previous urethral sling, artificial urinary sphincter, or penile prosthesis surgery.
* Any contraindication to MRI (contrast allergy, severe claustrophobia, MRI-incompatible prosthesis, MRI-unsafe aneurysm clips)

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — a prostate gland must be present
Enrollment: 2 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Adverse event monitoring | up to 12 months post treatment
  adverse event data will be monitored and tabulated. The primary study endpoint will be achieved by the absence of any Grade 3 or higher adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Brisbane, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided